CLINICAL TRIAL: NCT02333877
Title: Comparison of Skinlink With Suture for ED Patients: a Randomized Controlled Trial
Brief Title: Comparison of Skinlink With Suture for ED Patients
Acronym: Skinlink
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Kim Hyeongtae, Residency, Hallym University Kangnam Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Skinlink_SHH
Record Dates: First submitted 2015-01-04; First posted 2015-01-07 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Wounds and Injuries; Lacerations
MeSH Terms: conditions — Wounds and Injuries; Lacerations | interventions — Nylons

ARMS (2):
- Skinlink (Experimental): applying Skinlink on simple laceration (length < 5cm)
  Interventions: Other: Skinlink
- Nylon (Other): applying conventional suture using nylon on simple laceration (length < 5cm)
  Interventions: Other: Nylon

INTERVENTIONS:
Other: Skinlink — suture using Skinlink
  Arms: Skinlink
Other: Nylon — conventional suture using nylon
  Arms: Nylon

SUMMARY:
The purpose of this study is to determine whether suture using the Device of "Leukosan Skinlink" is more faster and safer than that of "nylon" in the treatment of simple wound for ED patients.

ELIGIBILITY:
The inclusion criteria were age 18-75 years,presence of a partial thickness laceration, generally good health without systemic abnormalities,agreement to return for a 14-day follow-up, and written informed consent. The exclusion criteria were previous diagnosis of diabetes mellitus, peripheral vascular disease, or bleeding disorders; history of keloid formation or scar hypertrophy; and allergy to cyanoacrylate compounds or formaldehyde

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Time required to complete suture | 1year

SECONDARY OUTCOMES:
Dehiscence | 1year
Infection rate | 1year

CONTACTS AND LOCATIONS:
Locations (1):
- Kangnam Sacred Heart Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim H, Kim W, Kang GH, Jang YS, Choi HY, Kim JG, Kim IY, Kim M. Comparison of Leukosan SkinLink with surgical suture for traumatic laceration repair: A randomized controlled trial. Medicine (Baltimore). 2018 Jun;97(25):e10918. doi: 10.1097/MD.0000000000010918. PMID 29923977